CLINICAL TRIAL: NCT05567471
Title: Phase 3, Randomized, Multi-Centric, Open-labeled Study to Evaluate Immunogenicity and Safety of BBV154 Booster Dose in Participants Previously Vaccinated With EUA Vaccines
Brief Title: Phase 3 Study to Evaluate Immunogenicity and Safety of BBV154 Booster Dose
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Bharat Biotech International Limited (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: BBIL/Booster/2021 Hetero
Record Dates: First submitted 2022-09-29; First posted 2022-10-05 (Actual); Last update posted 2022-10-05 (Actual); Status verified 2022-10

CONDITIONS: COVID-19 Respiratory Infection
MeSH Terms: interventions — ChAdOx1 nCoV-19

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- Group 1(BBV154 in COVAXIN recipients) (Active Comparator): 250 participants will be recruited and administered with a booster dose of BBV154 vaccine in form of drops (0.5 mL) via intranasal route, in individuals previously vaccinated with COVAXIN.
  Interventions: Biological: BBV154 Intranasal Vaccine
- Group 2 (COVAXIN in COVAXIN recipients) (Active Comparator): 125 participants will be recruited and administered with a booster dose of BBV152 vaccine, in individuals previously vaccinated with COVAXIN.
  Interventions: Biological: Intramuscular vaccine COVAXIN
- Group 3 (BBV154 in COVISHIELD recipients) (Active Comparator): 250 participants will be recruited and administered with a booster dose of BBV154 vaccine, in individuals previously vaccinated with COVISHIELD.
  Interventions: Biological: BBV154 Intranasal Vaccine
- Group 4(COVAXIN in COVISHIELD recipients) (Active Comparator): 125 participants will be recruited and administered with a booster dose of BBV152 (COVAXIN) vaccine, in individuals previously vaccinated with COVISHIELD.
  Interventions: Biological: Intramuscular vaccine COVAXIN
- Group 5 (COVISHIELD in COVISHIELD recipients) (Active Comparator): 125 participants will be recruited and administered with a booster dose of Covishield vaccine, in individuals previously vaccinated with COVISHIELD.
  Interventions: Biological: Covishield

INTERVENTIONS:
Biological: BBV154 Intranasal Vaccine — Administered BBV154 vaccine in form of drops (0.5 mL) via intranasal route
  Arms: Group 1(BBV154 in COVAXIN recipients); Group 3 (BBV154 in COVISHIELD recipients)
Biological: Intramuscular vaccine COVAXIN — Administered BBV152 vaccine via intramuscular route
  Arms: Group 2 (COVAXIN in COVAXIN recipients); Group 4(COVAXIN in COVISHIELD recipients)
Biological: Covishield — Administered vaccine via intramuscular route
  Arms: Group 5 (COVISHIELD in COVISHIELD recipients)

SUMMARY:
A total sample size of 875 healthy volunteers ages ≥18 years will be recruited in this study in the ratio of 2:1:2:1:1.

Group 1: (BBV154 in COVAXIN recipients): In this group, 250 participants will be recruited and administered with a booster dose of BBV154 vaccine in form of drops (0.5 mL) via intranasal route, in individuals previously vaccinated with COVAXIN.

Group 2: (BBV152(COVAXIN) in COVAXIN recipients): In this group, 125 participants will be recruited and administered with a booster dose of BBV152 vaccine, in individuals previously vaccinated with COVAXIN.

Group 3: (BBV154 in COVISHIELD recipients) In this group, 250 participants will be recruited and administered with a booster dose of BBV154 vaccine, in individuals previously vaccinated with COVISHIELD.

Group 4: (BBV152(COVAXIN) in COVISHIELD recipients) In this group, 125 participants will be recruited and administered with a booster dose of BBV152 (COVAXIN) vaccine, in individuals previously vaccinated with COVISHIELD.

Group 5: (COVISHIELD in COVISHIELD recipients) In this group, 125 participants will be recruited and administered with a booster dose of Covishield vaccine, in individuals previously vaccinated with COVISHIELD.

DETAILED DESCRIPTION:
Sample Collection:

1. Pregnancy test will be conducted by using rapid test kit throughout the study.
2. Immunogenicity analysis: A total of 5 ml of blood is collected at days 0, 28, 56 (Subset n=150 each in Groups 1 &3 and 75 each in Groups 2, 4, and 5). Sera will collect from the blood sample and stored as 3 aliquots at -20°C.
3. An additional blood sample (10 mL) will be collected for assessment of cell mediated responses on days 0, 28, 56 (Subset n=40each in Groups 1 & 3 and 20 each in Groups 2, 4, and 5).
4. A saliva sample (5 mL) will be collected on days 0, 28, 56 (Same subset as for assessment of cell mediated responses). Saliva will be collected by Passive drool method using Falcon tube.

Sample Size:

A total sample size of 875 healthy volunteers ages ≥18 years will be recruited in this study

Randomization:

A total sample size of 875 healthy volunteers ages ≥18 years will be recruited in this study in the ratio of 2:1:2:1:1.

Block randomization with an integrated web response will be utilized to ensure balance among the four groups, with a 2:1:2:1:1 ratio allocation of Group 1, 2, 3, 4 and 5 respectively.

STUDY RATIONALE:

The reasons for booster doses may differ by population groups at risk, type of vaccine, waning immunity, variants of concern, and clinical and epidemiological settings (1). Studies have shown that immunity after vaccination against SARS-CoV-2 infection wanes in a few months of time, which suggests the need for a booster dose. The emergence of SARS-CoV-2 variants due to multiple mutations in the Spike protein, such as Delta (B.1.617.2) variant in India and Beta strain (B.1.351) in South Africa have raised concerns because of their increased transmission rates.

As and when other variants emerge that are going to be worse than the present Covid-19 variants and has the potency to evade the currently available vaccines, then the requirement of booster shots would be needed. The most recent data from Israel and the United States in the context of the delta Variant of Concern (VOC) predominant circulation suggest that vaccine protection against COVID-19 infection wanes approximately 6 to 8 months following the second dose . Emory University, USA has been published the data that shown a 7 fold reduction in the antibody titer against SARS-CoV-2 virus in a span of 6 months post-vaccination with mRNA vaccine . The CDC, USA recommended the booster dose the individuals who are moderately to severely immunocompromised and not able to build enough protection in the first vaccination .

Globally, many countries like Israel, the UAE, Russia, France, Germany and Italy have already rolled out boosters. In Israel, where the country began offering boosters to people over 60 in July, early data suggests that a Pfizer booster dose can significantly improve immunity among people in that age group. The booster dose, the data indicated, reduced risk of infection in people 60 and were about 19.5 times less likely to have severe COVID-19 than were people in the same age group who had received only two jabs and were studied during a similar time period .

Study Design:

The Phase-III study is designed to evaluate the immunogenicity and safety of volunteers who receive either BBV154 vaccine via intranasal route or BBV152 vaccine via intramuscular route or COVISHIELD via intramuscular route when administered as booster dose in individuals previously vaccinated with EUA vaccines in India .A total of 875 participants will be enrolled, randomized and will be conducted in open labeled manner.

Group 1 (BBV154 in COVAXIN recipients): In this group, 250 participants will be recruited and administered with a booster dose of BBV154 vaccine in form of drops (0.5 mL) via intranasal route, in individuals previously vaccinated with COVAXIN.

Group 2 (BBV152 in COVAXIN recipients): In this group, 125 participants will be recruited and administered with a booster dose of BBV152 vaccine, in individuals previously vaccinated with COVAXIN.

Group 3 (BBV154 in COVISHIELD recipients) In this group, 250 participants will be recruited and administered with a booster dose of BBV154 vaccine via intranasal route, in individuals previously vaccinated with COVISHIELD.

Group 4 (BBV152 in COVISHIELD recipients) In this group, 125 participants will be recruited and administered with a booster dose of BBV152 vaccine, in individuals previously vaccinated with COVISHIELD.

Group 5 (COVISHIELD in COVISHIELD recipients) ) In this group, 125 participants will be recruited and administered with a booster dose of Covishield vaccine, in individuals previously vaccinated with COVISHIELD.

In addition to administering the vaccine, a series of blood samples (Immunogenicity Subset) will be collected for analyzing serum for immunological assessments.

A subset of 150 participants each in Groups 1 &3 and 75 participants each in Groups 2, 4, and 5 will be assessed for immunogenicity. Among this subset an additional 10 mL blood and 5 mL of saliva will be collected from 40 participants each in Groups 1 &3 and 20 participants each in Groups 2, 4, and 5 to assess the cell-mediated immune response and mucosal immunity, respectively.

STUDY PROCEDURES:-

Visit 1: Baseline (Day 0):

1. The participant will be screened for eligibility based on medical history, vitals, and physical examination.
2. If the participant is eligible (in good general health or stable pre-existing disease as per the discretion of the Principal investigator), a blood sample will be withdrawn prior to vaccination for all the participants.
3. Blood sample (5 mL) will be collected from the subset of participants (n=150 each in Groups 1 &3 and n=75 each in Groups 2, 4, and 5).
4. 5 mL saliva and additional blood sample (10 mL for PBMC) will be collected to assess the secretary IgA Ab titer and cell mediated immune response in subset (n=40 in groups 1&3 and n=20 in groups2,4,5).
5. A study vaccine will be administered. Following vaccination, participants will remain at the study site for at least 30 minutes of observation to record any immediate adverse event.
6. Diary card will be distributed to the participants.
7. Telephonic follow-up at 15 ± 2 days intervals for assessing health status, and general and COVID-19 symptoms history.

Visit 2 (Day 28 + 2 days):

1. Study participants will return to the OPD for vitals and physical examination (general and systemic examination), and specific symptoms for COVID-19.
2. For the humoral immunogenicity subset, 5mL of blood will be collected and processed for serum for assessing neutralizing responses (150 each in Groups 1 &3 and n=75 each in Groups 2, 4, and 5).
3. 5 mL saliva and additional blood sample (10 mL for PBMC) will be collected to assess the secretary IgA Ab titer and cell mediated immune response in subset (n=40 in groups 1&3 and n=20 in groups2,4,5)
4. Telephonic follow-up for all the other participants at 15±2 days intervals for assessing health status, and general and COVID-19 symptoms history.

Visit 3 (Day 56 ± 7 days):

1. Study participants will return to the OPD for physical examination (general and systemic examination), and specific symptoms for COVID-19.
2. For the humoral immunogenicity subset, 5mL of blood will be collected and processed for serum for assessing neutralizing responses (150 each in Groups 1 &3 and n=75 each in Groups 2, 4, and 5).
3. 5 mL saliva and additional blood sample (10 mL for PBMC) will be collected to assess the secretary IgA Ab titer and cell mediated immune response in subset (n=40 in groups 1&3 and n=20 in groups2,4,5)
4. Telephonic follow-up for all the other participants at 15±2 days intervals for assessing health status, and general and COVID-19 symptoms history.

Visit 4 (Day 90± 7 days):

Telephonic follow-up for all the other participants for assessing health status, and general and COVID-19 symptoms history.

Visit 5 (Day 180 ± 7 days):

Telephonic follow-up for all the other participants for assessing health status, and general and COVID-19 symptoms history

Safety Monitoring:

Subjects will be observed for 30 minutes after vaccination for immediate adverse events. Active surveillance will be conducted for all participants for seven days after vaccination to ascertain information on solicited adverse events ("Reactogenicity").

ELIGIBILITY:
Inclusion Criteria:

1. Ability to provide written informed consent.
2. Participants of either gender of age ≥18 years.
3. Received and completed COVID-19 vaccine under Emergency Use Authorization (EUA) dosing guidelines at least 6 ± 1 month (after receipt of second dose of EUA vaccine) prior to enrollment, confirmed by the electronic Covid-19 Certificate (CoWIN).
4. Expressed interest and availability to fulfill the study requirements.
5. For a female participant of child-bearing potential, planning to avoid becoming pregnant (use of an effective method of contraception or abstinence) from the time of study enrolment until at least four weeks after the vaccination.
6. Agrees not to participate in another clinical trial at any time during the study period.
7. Agrees to remain in the study area for the entire duration of the study.
8. Willing to allow storage and future use of biological samples for future research

Exclusion Criteria:

1. Known history of COVID-19 infection.
2. For women of child bearing potential, a positive serum pregnancy test (during screening within 45 days of enrolment) or positive urine pregnancy test (within 24 hours of administering of vaccine).
3. Temperature >38.0°C (100.4°F) or symptoms of an acute self limiting illness such as an upper respiratory infection or gastroenteritis within three days prior to vaccination.
4. Medical problems because of alcohol or illicit drug use during the past 12 months.
5. Receipt of an experimental agent (vaccine, drug, device, etc.) within 60 days before enrolment or expects to receive an investigational agent during the study period.
6. Receipt of any licensed vaccine within four weeks before enrolment in this study.
7. Known sensitivity to any ingredient of the study vaccines, or a more severe allergic reaction and history of allergies in the past.
8. Receipt of immunoglobulin or other blood products within the three months prior to vaccination in this study.
9. Immunosuppression because of an underlying illness or treatment with immunosuppressive or cytotoxic drugs or use of anticancer chemotherapy or radiation therapy within the preceding 36 months.
10. Long-term use (> 2 weeks) of oral or parenteral steroids (glucocorticoids) or high dose inhaled steroids (>800 mcg/day of beclomethasone dipropionate or equivalent) within the preceding six months (nasal and topical steroids are allowed).
11. Any history of anaphylaxis in relation to vaccination.
12. History of any cancer.
13. History of severe psychiatric conditions likely to affect participation in the study.
14. A bleeding disorder (e.g. factor deficiency, coagulopathy or platelet disorder, or prior history of significant bleeding or bruising following IM injections or venepuncture).
15. Any other serious chronic illness requiring immediate hospital specialist supervision.
16. Any other condition that in the opinion of the investigator would jeopardize the safety or rights of a volunteer participating in the trial or would render the subject unable to comply with the protocol.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 875 (Actual)
Dates: Start 2022-02-26 (Actual); Primary Completion 2022-05-03 (Actual); Study Completion 2022-09-28 (Actual)

PRIMARY OUTCOMES:
Geometric mean titres 1 | baseline
  Serum neutralising antibody titer (NAb"s) by neutralizing antibody assays.
Geometric mean titres 2 | Day 28+2
  Serum neutralising antibody titer (NAb"s) by neutralizing antibody assays.
Geometric mean titres 3 | Day 56 ± 7
  Serum neutralising antibody titer (NAb"s) by neutralizing antibody assays.

SECONDARY OUTCOMES:
Geometric mean titres 4 | Day 28+2
  GMTs of serum IgG Abs by ELISA
Geometric mean titres 5 | Day 56 ± 7
  GMTs of serum IgA Abs by ELISA
Cell mediated immune response | Day 28+2
  Vaccine induced T cell responses through cell mediated immune analysis
Cell mediated immune response | Day 56 ± 7
  Vaccine induced B cell responses through cell mediated immune analysis
Geometric mean titres | Day 28+2
  GMTs of secretary IgA Abs by ELISA.
Geometric mean titres (GMTs) | Day 56 ± 7
  GMTs of secretary IgA Abs by ELISA.
adverse events reported | 7 days after vaccination
  The occurrence of solicited adverse events
adverse events of special interest reported | throughout the study duration 7 months
  The occurrence of adverse event of special interest (AESI).
vaccine induced thrombosis and thrombocytopenia | throughout the study duration 7 months
  The occurrence of the vaccine induced thrombosis and thrombocytopenia in participants reporting the respective symptoms and signs.

CONTACTS AND LOCATIONS:
Overall Officials: Dr. Sanjay Rai, MBBS,MD, Principal Investigator — AIIMS, New Delhi; Dr Chandramani Singh, MBBS,MD, Principal Investigator — All India Institute of Medical Sciences; Dr Anil Kumar Pandey, MBBS,MD, Principal Investigator — ESIC Medical College and Hospital Faridabad; Dr Chandrashekhar S Gillurkar, MBBS,MD, Principal Investigator — Gillurkar Multispeciality Hopistal; Dr Amit Suresh Bhate, MBBS,MD, Principal Investigator — Jeevan Rekha Hospital; Dr Jitendra Singh Kushwaha, MBBS,MD, Principal Investigator — Prakhar Hospital Pvt Ltd; Dr Shivaraj K K, MBBS,MD, Principal Investigator — Vagus Super Specilaity Hospitals; Dr A Venkateshwar Rao, MBBS,MD, Principal Investigator — St. Theresa Hospital; Dr Ajeet Pratap Singh, MBBS,MD, Principal Investigator — Rana Hospital Pvt Ltd
Locations (9):
- India (9):
  - All India Institute of Medical Sciences, Patna, Bihar
  - ESIC Medical College and Hospital, Faridabad, Haryana
  - Vagus Super Specilaity Hospitals, Bangalore, Karnataka
  - Jeevan Rekha Hospital, Belagavi, Karnataka
  - Gillurkar Multispeciality Hopistal, Nagpur, Maharashtra
  - St. Theresa Hospital, Hyderabad, Telangana
  - Rana Hospital Pvt Ltd, Gorakhpur, Uttar Pradesh
  - Prakhar Hospital Pvt Ltd, Kanpur, Uttar Pradesh
  - AIIMS, New Delhi, New Delhi